CLINICAL TRIAL: NCT05534243
Title: Awareness With Paralysis and Post-Traumatic Stress Disorder Among Mechanically Ventilated Emergency Department Survivors: the ED-AWARENESS-2 Trial
Brief Title: The ED-AWARENESS-2 Trial
Acronym: ED-AWARENES II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Brian Fuller, Associate Professor of Anesthesiology (Critical Care Medicine) and Emergency Medicine, Washington University School of Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202207132; 1R01HL162721-01A1 (NIH)
Record Dates: First submitted 2022-09-02; First posted 2022-09-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-02

CONDITIONS: Awareness; Mechanical Ventilation; Intubation Complication; PTSD
Keywords: Awareness; Paralysis; Emergancy Department; Rocuronium; Mechanical Ventilation; Intubation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Paralysis | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Multicenter, stepped wedge, cluster randomized trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Before group (Active Comparator): Mechanically ventilated emergency department patients receiving standard neuromuscular blockers prior to an educational initiative on the importance of ED-based targeted shorter acting neuromuscular blocker.
  Interventions: Other: Standard neuromuscular blocker practices
- After group (Experimental): Mechanically ventilated emergency department patients receiving neuromuscular blockers after an educational initiative aimed at improving use of shorter acting neuromuscular blocker practices in the ED.
  Interventions: Behavioral: Education

INTERVENTIONS:
Other: Standard neuromuscular blocker practices — Usual care neuromuscular blocker in the ED
  Arms: Before group
Behavioral: Education — Nurses and physicians will be engaged regarding the clinical outcome data on the importance of shorter acting neuromuscular blockers, and the objectives of the research. Education will include in-services and lectures focused on the importance of neuromuscular blocker protocols on patient outcome. The use of neuromuscular blokers will be evaluated throughout the study in order to better understand providers' perception of and experience with ED-based neuromuscular blocker protocols.
  Arms: After group

SUMMARY:
The investigators will screen all mechanically ventilated ED patients for study eligibility and will enroll all consecutive patients satisfying inclusion and exclusion criteria.

The study design is a pragmatic, multicenter, stepped wedge cluster randomized trial, enrolling at five sites over a 3-year period, divided into six time periods of six months. Prior to the study, each site will be randomized to their position within the design. One site will cross to the intervention period (i.e. succinylcholine as default neuromuscular blocker) every six months from the 2nd to 6th time period. Cluster order will be determined by computer-based randomization. To begin, each site will be exposed to control conditions; by the end of the study, each site will be exposed to intervention conditions.

Patients in the control phase will receive usual care, and this phase will be entirely observational. After six months, a site will enter a 2-month transition phase. In this phase, the investigators will implement the intervention, similar to how they have implemented other ED-based interventions for mechanically ventilated patients. The investigators will engage and educate ED clinicians on the importance of AWP prevention and the study objectives. The intervention framework relies on the use of "nudges", without restricting choice. The use of neuromuscular blockers (i.e. "paralytic" medications) is already part of routine care in the ED in order to facilitate endotracheal intubation and initiation of mechanical ventilation for patients with acute respiratory failure. The two most common neuromuscular blockers used in the ED are succinylcholine and rocuronium. The preliminary data show a strong association between rocuronium (a longer-acting neuromuscular blocker) use and AWP. Therefore, this study aims to improve care by educating caregivers on AWP and the use of the neuromuscular blockers, which are already routinely used, and studying that process in a rigorous fashion. The default neuromuscular blocker in the intervention phase will be succinylcholine. Succinylcholine will be the default over rocuronium because: 1) it has safely been the default neuromuscular blocker of choice in the ED for >40 years ; 2) its 5-minute duration of action greatly reduces AWP risk; 3) the preliminary data regarding an increased risk of AWP with rocuronium and 4) ED rocuronium use has increased despite no patient-centered studies showing benefit over succinylcholine. Passive alerts (i.e. graphics, pocket cards) will also be strategically placed in the ED, and active alerts will be used as reminders before every nursing shift (i.e. "the huddle"). After this transition phase, the site will begin the intervention phase, and patients will again receive clinician-directed care, just after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanical ventilation via an endotracheal tube
2. Age ≥ 18 years
3. Treatment with a neuromuscular blocker (for endotracheal intubation or during the post-intubation phase of care)

Exclusion Criteria:

1. Acute or chronic neurologic injury with deficit that prevents assessment of AWP (i.e. stroke, intracranial hemorrhage, traumatic brain injury, cardiac arrest, severe dementia)
2. Death before extubation
3. Transfer to another hospital from the ED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3090 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
The prevention of Awareness with Paralysis, as assessed by the modified Brice questionnaire. | up to 30 days
  The modified Brice questionnaire will be used in this trial.

SECONDARY OUTCOMES:
PTSD symptoms | 30 days
  Will be measured using the PCL-5, a validated 20-item (score 0-4, Likert scale) self-reported measure that assesses 20 DSM-5 symptoms of PTSD.
PTSD symptoms | 180 days
  Will be measured using the PCL-5, a validated 20-item (score 0-4, Likert scale) self-reported measure that assesses 20 DSM-5 symptoms of PTSD.
Depression and Anxiety | 30 days
  Hospital Anxiety and Depression Scale (HADS), a validated 14-item (7 depression, 7 anxiety, ordinal score 0-3) questionnaire commonly used in critical illness
Depression and Anxiety | 180 days
  Hospital Anxiety and Depression Scale (HADS), a validated 14-item (7 depression, 7 anxiety, ordinal score 0-3) questionnaire commonly used in critical illness
Health Related Quality of Life (QOL) | 30 days
  EuroQol-5D (EQ-5D), the most widely used scale for measuring health-related QOL and part of the core sets recommended for critical care studies on post-discharge outcomes
Health Related Quality of Life (QOL) | 180 days
  EuroQol-5D (EQ-5D), the most widely used scale for measuring health-related QOL and part of the core sets recommended for critical care studies on post-discharge outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Brian Fuller, MD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Roy J. and Lucille A. Carver College of Medicine, Iowa City, Iowa
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Cooper University Hospital/Cooper Medical School of Rowan University, Camden, New Jersey
  - University of Washington School of Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
We will consider sharing IPD upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after all publications related to the data.
Access Criteria: Can be obtained by contacting the study PI.

REFERENCES:
- [Derived] Fuller BM, Driver BE, Roberts MB, Schorr CA, Thompson K, Faine B, Yeary J, Mohr NM, Pappal RD, Stephens RJ, Yan Y, Johnson NJ, Roberts BW. Awareness with paralysis and symptoms of post-traumatic stress disorder among mechanically ventilated emergency department survivors (ED-AWARENESS-2 Trial): study protocol for a pragmatic, multicenter, stepped wedge cluster randomized trial. Trials. 2023 Nov 25;24(1):753. doi: 10.1186/s13063-023-07764-5. PMID 38001507